CLINICAL TRIAL: NCT05676216
Title: Efficacy of Sodium Bicarbonate for Treatment of Acute Peripheral Vertigo: A Double-blinded Randomized Control Trial
Brief Title: Sodium Bicarbonate for Acute Peripheral Vertigo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202209092MIND
Record Dates: First submitted 2022-12-12; First posted 2023-01-09 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2022-12

CONDITIONS: Peripheral Vertigo
Keywords: Sodium Bicarbonate; Diphenhydramine
MeSH Terms: conditions — Vertigo | interventions — Diphenhydramine; Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Diphenhydramine (Active Comparator): Diphenhydramine 30 mg in 100 mL normal saline intravenous dripping
  Interventions: Drug: Diphenhydramine
- Sodium Bicarbonate (Experimental): Sodium bicarbonate 66.4 mEq in 100 mL normal saline intravenous dripping
  Interventions: Drug: Sodium Bicarbonate
- Diphenhydramine with Sodium Bicarbonate (Experimental): Diphenhydramine 30 mg in 100 mL normal saline intravenous dripping with Sodium bicarbonate 66.4 mEq intravenous push
  Interventions: Drug: Diphenhydramine + Sodium Bicarbonate

INTERVENTIONS:
Drug: Diphenhydramine — Diphenhydramine 30 mg in 100 mL normal saline intravenous dripping when vertigo patients visit Emergency Department
  Arms: Diphenhydramine
Drug: Sodium Bicarbonate — Sodium bicarbonate 66.4 mEq in 100 mL normal saline intravenous dripping when vertigo patients visit Emergency Department
  Arms: Sodium Bicarbonate
Drug: Diphenhydramine + Sodium Bicarbonate — Diphenhydramine 30 mg in 100 mL normal saline intravenous dripping with Sodium bicarbonate 66.4 mEq intravenous push when vertigo patients visit Emergency Department
  Arms: Diphenhydramine with Sodium Bicarbonate

SUMMARY:
Vertigo is defined as the hallucination of spinning sensation or rotatory movement and is frequently combined with severe nausea and vomiting. In Taiwan, an average of 3.13 cases per 100 persons suffer from acute vertigo attack per year. And 1 in 3 patients with vertigo will have recurrent attack within a year. The sensation of disequilibrium and severe nausea and vomiting urge patients visit emergent department (ED) for help. Therefore, vertigo is one of the most common complaints in ED.

Vertigo can be divided into central type and peripheral type. Central type vertigo included life threatening disease like brainstem hemorrhage or infraction. Although peripheral vertigo is mostly benign, the acute symptoms relief are usually needed. The first line therapy of acute peripheral vertigo is using antihistamine or benzodiazepine with other anti-emetic agents. However, these agents usually have side effects of fatigue and lethargy, which will cause increasing patients' length of stay or elders' risk of falling.

Sodium bicarbonate is widely used in treating hyperkalemia or metabolic acidosis. Its safety and no side effect have also been proved. There were few reports of using sodium for treatment of acute vertigo in Taiwan and Japan. However, there is no strong evidence of comparing this therapy with other medication.

This study hypothesized that there is an equivalence of efficacy between sodium bicarbonate and diphenhydramine for treatment of vertigo. Using sodium can cause less fatigue or lethargy and can decrease ED length of stay. This study aims to perform a double-blinded randomized controlled trial to evaluate the efficacy of sodium bicarbonate for treatment of acute peripheral vertigo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute onset vertigo

Exclusion Criteria:

* Pregnancy
* First vertigo episode over 24 hours
* Using any anti-vertigo medicine after onset
* Drug allergy to Sodium bicarbonate or Diphenhydramine
* Diagnosed with central vertigo
* Heart failure NYHA class >1
* Chronic kidney disease (CKD) stage ≥ 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2023-01-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction in vertigo intensity | Baseline and 60 minutes after drug administration
  Reduction in Vertigo Visual Analog Scale (VAS 0~10, higher scores mean higher intensity) from baseline

SECONDARY OUTCOMES:
Reduction in nausea intensity | Baseline and 60 minutes after drug administration
  Reduction in Nausea Visual Analog Scale (VAS 0~10, higher scores mean higher intensity) from baseline
Improvement of ambulatory ability | Baseline and 60 minutes after drug administration
  Change in objective ambulatory ability (score 1~4, higher scores mean a worse outcome) from baseline
Lethargy | 60 minutes after drug administration
  Lethargy score (score 1~4, 1 indicates no lethargy and 4 indicates very lethargy)
Emergency Department staying time | up to 24 hours
  From patients admit to Emergency Department until patients discharge (up to 24 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Yu Chi, MD, Principal Investigator — Emergency Department, National Taiwan University, Yunlin Branch
Locations (1):
- National Taiwan University Yunlin Branch, Yunlin County, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hunter BR, Wang AZ, Bucca AW, Musey PI Jr, Strachan CC, Roumpf SK, Propst SL, Croft A, Menard LM, Kirschner JM. Efficacy of Benzodiazepines or Antihistamines for Patients With Acute Vertigo: A Systematic Review and Meta-analysis. JAMA Neurol. 2022 Sep 1;79(9):846-855. doi: 10.1001/jamaneurol.2022.1858. PMID 35849408
- [Background] Numata K, Shiga T, Omura K, Umibe A, Hiraoka E, Yamanaka S, Azuma H, Yamada Y, Kobayashi D. Comparison of acute vertigo diagnosis and treatment practices between otolaryngologists and non-otolaryngologists: A multicenter scenario-based survey. PLoS One. 2019 Mar 7;14(3):e0213196. doi: 10.1371/journal.pone.0213196. eCollection 2019. PMID 30845218
- [Derived] Chi CY, Chen YC, Cheng MT, Chang KC, Chen YP, Tsai MS, Chang WT, Ma MH, Huang CH, Chiang WC. Diphenhydramine, Sodium Bicarbonate, or Combination for Acute Peripheral Vertigo: A Randomized Clinical Trial. JAMA Netw Open. 2025 Nov 3;8(11):e2541472. doi: 10.1001/jamanetworkopen.2025.41472. PMID 41196596